CLINICAL TRIAL: NCT01060943
Title: A Randomized, Multicenter, Prospective, Paired Comparison of the Efficacy and Safety of TheraFill® Versus KOKEN for 3 Months on Nasolabial Folds
Brief Title: An Efficacy and Safety Study of TheraFill® Versus KOKEN for 3 Months on Nasolabial Folds
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sewon Cellontech Co., Ltd. (Industry)
Responsible Party: Jong Won, Lee, Kangnam St.Mary's Hospital of Catholic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01TRF
Record Dates: First submitted 2010-01-21; First posted 2010-02-02 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-02

CONDITIONS: Nasolabial Folds
Keywords: injectable collagen filler; correction of wrinkles and folds; enrolled : 73; withdrawal : 4; ongoing : 0; completed : 69

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KOKEN(collagen) (Active Comparator): atelocollagen filler
  Interventions: Device: KOKEN
- TheraFill (Experimental): atelocollagen filler
  Interventions: Device: Atelocollagen Filler

INTERVENTIONS:
Device: KOKEN — atelocollagen filler
  1ml pre-filled syringe. 3% atelocollagen is dissolved in PBS. Inject several times every 2 weeks or more weeks. Total amount should be limited up to 25ml per an year.
  Other Names: KOKEN ATELOCOLLAGEN FILLER
  Arms: KOKEN(collagen)
Device: Atelocollagen Filler — 1ml pre-filled syringe. 3% atelocollagen is dissolved in PBS. Inject several times every 2 weeks or more weeks. Total amount should be limited up to 25ml per an year.
  Other Names: TheraFill ATELOCOLLAGEN FILLER
  Arms: TheraFill

SUMMARY:
* Investigational Device : TheraFill® (Atelocollagen Dermal Filler)
* Title : A Randomized, Multicenter, Prospective and Paired Comparison of the Efficacy and Safety of TheraFill® versus KOKEN for 3months on Nasolabial Folds
* Sites and investigators :

  * The Catholic University of Korea. Kangnam St. Mary's Hospital (#505, Banpo-dong, Seocho-gu, SEOUL)
  * The Catholic Univ. of Korea Holy Family Hospital (#2, Sosa-dong, Wonmi-gu, Bucheon-si, Gyeonggi-do)
* Objective : To compare the non-inferiority of TheraFill® with KOKEN for evaluation of the efficacy and safety on Nasolabial Folds for 3months
* Clinical Study Method : Seventy-three subjects who agree to voluntarily participate in the clinical study are randomized to treatment with TheraFill (porcine atelocollagen filler) and KOKEN (bovine atelocollagen filler) in the contralateral fold(NFL). The subjects shall regularly visit the hospital 5 times or more and if subjects take touch-up treatments, the number of visit times will be increased. Treatments shall be repeated at 2 weeks intervals, as required, to achieve "Optimal cosmetic result". Outcomes shall be evaluated by blinded investigators, investigators and subjects at 2,4 and 12 weeks after baseline.
* Subjects : The target number of subjects is 62subjects, and 73 subjects are selected in the screening period in consideration of 15% of dropout rate.

DETAILED DESCRIPTION:
* Evaluation Criteria And Analysis Method :

  1. Efficacy - Evaluate total 3 times : 2, 4 and 12 weeks after last injection. In efficacy evaluation data, for difference in WSRS improvement ratio, normality test on the ratio is used, and for the other evaluation variables, statistical hypothesis test is conducted by using t-test, Wilcoxon rank-sum test, Chi-square test, and ANOVA for repeatedly measured data according to the nature of data.
  1. Wrinkle Severity Rating System - It is ranged from 1 point (absent) to 5 points (extreme), and WSRS scores are compared baseline(pre-injection period) with every visits.
  2. Evaluation of subject's improvement - It is ranged from 1 point (worse) to 5 points (much improved). A degree of improvement to which the subject decides upon every visit is evaluated, compared to the screening period (baseline).
  3. Evaluation of investigator's improvement - It is ranged from 1 point (worse) to 5 points (much improved). A degree of improvement to which the investigator decides upon every visit is evaluated, compared to the screening period (baseline).

  2. Safety The analysis of safety evaluation data is conducted through descriptive statistics using the causal relationship between outbreak frequency and the devices .
  1. Subjective adverse events : Uncomfortable sense after TheraFill® injection
  2. Objective adverse events : Investigator shall observe and evaluate adverse events such as edema, redness, tenderness, pain, bruise, itching, nodule and others at injected site after injection
* Evidence : 1. Photographs At screening period, injection, 2, 4 and 12 weeks after injection and upon an adverse event, the photograph results of the front and side shall be attached to the Case Report Form and utilized as objective reference data.

ELIGIBILITY:
Inclusion Criteria:

1. Those who agreed to this treatment and signed the Informed Consent Form
2. Those who are 20 years old or more and desire to take correction of nasolabial folds
3. Those who have an intention of refraining from other cosmetic treatment(other filler injection, laser or chemical peeling, Botox injection or wrinkle reduction) during the clinical study period
4. Those whose Wrinkle Severity Rating Scale (WSRS) is more than 2 points at least

Exclusion Criteria:

1. Subjects or their families who currently have or have the history of autoimmune disease or collagen vascular disease
2. Those who had the history of anaphylactic response
3. Those who are sensitive to implant
4. Those who are sensitive to lidocaine or other amide anesthesia
5. Those who are sensitive to porcine protein
6. Those who are sensitive to control device
7. Those who have taken soft tissue augmentation, laser or cosmetic facial surgery to improve the injection area in 6 months before participation in the clinical study
8. Those who are pregnant or lactating, or expect pregnancy
9. Those who have inflammatory skin disease on the injection area
10. Those who are judged by the subinvestigator to be improper for this study due to mental disease etc.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Efficacy: Wrinkle Severity Rating Scale - Primary endpoint | At screening period, 2, 4 and 12 weeks after last injection
Efficacy: An assessment of the degree of improvement based on the judgement of patients | At screening period, 2, 4 and 12 weeks after last injection
Efficacy: An assessment of the degree of improvement based on the judgement of the Investigators | At screening period, 2, 4 and 12 weeks after last injection

CONTACTS AND LOCATIONS:
Overall Officials: Jong Won Lee, Ph.D, Principal Investigator — St.Mary's Hospital of Catholic University
Locations (1):
- Kangnam St.Mary's Hospital of Catholic University, Seoul, Seo-cho, South Korea